CLINICAL TRIAL: NCT03063281
Title: Association Between the Presence of Autoantibodies Targeting Ficolin-2 and Active Nephritis in Patients With Systemic Lupus Erythematosus
Brief Title: Anti-ficolin-2 Autoantibodies in Lupus Nephritis
Acronym: Ficolupus2
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Hospital, Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2030950v0
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: ficolin-2; anti-ficolin-2 antibodies; lupus nephritis; Lupus Erythematosus, Systemic; biomarker; ficolin-3; anti-ficolin-3 antibodies
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — Biological Oxygen Demand Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — one serum per patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SLE patient: 165 SLE patients. Subgroup : 77 with active lupus and 88 in disease remission. in the active subgroup : 36 with lupus nephritis and 41 without. Biological analysis were performed.
  Interventions: Other: BIological analysis
- healthy patients: 48 healthy patients. Biological analysis were performed.
  Interventions: Other: BIological analysis

INTERVENTIONS:
Other: BIological analysis — Biological analysis : ficolin-2 et anti-ficolin-2 antibodies
  Other Names: Biological analysis on preexisting

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disease characterized by the production of multiple autoantibodies. The prevalence and significance of antibodies against Ficolin-2 have not been yet investigated. The aims of this study were to determine the prevalence of anti-ficolin-2 antibodies among SLE patients and to investigate their potential as diagnostic and/or prognostic biomarkers in SLE.

This study is a secondary phase of a serum sample analysis done in early 2015 in order to determine the prevalence of anti-ficolin-2 antibodies among the same cohort as the previously declared study (ClinicalTrials.gov ID: NCT02625831; Unique Protocol ID: 1841851v0).

In this retrospective study, clinical data were obtained from medical files and blood samples were selected from preexisting biological collection. SLE patients (n=165) were informed and did not objected, they were matched to healthy controls (n=48). Disease activity was determined according to the SLEDAI score. Anti-ficolin-2 antibodies levels were measured in sera by ELISA and correlated to previously obtained Anti-ficolin-3, Anti-ficolin-2, anti-dsDNA and anti-C1q antibodies levels.

The titer of anti-ficolin-2 antibodies was correlated with the SLEDAI score (p<0.0001). The presence of anti-ficolin-2 antibodies was associated with anti-ficolin-3 antibodies, anti-C1q and anti-dsDNA antibodies.

Interestingly, the combination of anti-ficolin-3, anti-ficolin-2 and anti-C1q antibodies demonstrated higher specificity than any other traditional biomarker.

These results suggest that anti-ficolin-3 and anti-ficolin-2 antibodies could be useful for the diagnosis of active nephritis in SLE patients.

DETAILED DESCRIPTION:
For this retrospective study, the well written brief summary should be sufficient.

ELIGIBILITY:
165 SLE patients

Inclusion Criteria:

* Age: ≥ 18 years old
* Patients with lupus diagnostic criteria (ACR1997)

Exclusion Criteria:

* Pregnant women
* Patient with known evolutive cancer

  48 healthy patients matched in age and sex with one or several SLE patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SLE patients were studied from medical data files of the Departments of Internal Medicine (Grenoble University Hospital, France) and Nephrology (Conception University Hospital, Marseille, France). For SLE patients, clinical and biological manifestations as well as treatments received and disease activity evaluated using the SLE Disease Activity Index (SLEDAI) at the time of sampling were recorded. SLE patients were divided into subgroups as described in group section.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Anti-ficolin-2 antibodies presence in SLE patients | measured at day of inclusion = T0
  Anti-ficolin-2 antibodies in SLE patients, considered positive if superior than 95 arbitrary units.
  This study have a single visit approach with serum collection so every outcome is measured at T0, which is the only visit for the patient.

SECONDARY OUTCOMES:
Correlation of anti-ficolin-2 antibodies with anti-DNA antibodies in SLE patients | measured at day of inclusion = T0
  Correlation between Anti-ficolin-2 antibodies presence and anti-DNA antibodies presence.
  This study have a single visit approach with serum collection so every outcome is measured at T0, which is the only visit for the patient.
Correlation of anti-ficolin-2 antibodies with anti-C1q antibodies in SLE patients | measured at day of inclusion = T0
  Correlation between Anti-ficolin-2 antibodies presence and anti-C1q antibodies presence.
  This study have a single visit approach with serum collection so every outcome is measured at T0, which is the only visit for the patient.
Correlation of anti-ficolin-2 antibodies with lupus activity (SLEDAI score) in SLE | measured at day of inclusion = T0
  Correlation between Anti-ficolin-2 antibodies presence and clinical and/or biological evidence of SLE activity according to SLEDAI score (2012).
  This study have a single visit approach with serum collection so every outcome is measured at T0, which is the only visit for the patient.
Correlation of anti-ficolin-2 antibodies presence with active nephritis in SLE patients | measured at day of inclusion = T0
  Correlation between Anti-ficolin-2 antibodies presence and clinical and/or biological evidence of active nephritis This study have a single visit approach with serum collection so every outcome is measured at T0, which is the only visit for the patient.

IPD SHARING:
Plan to Share IPD: Undecided
Further analysis of serum collection is ongoing. IPD availability will be decided by the sponsor at completion and publication.

REFERENCES:
- [Background] Kuraya M, Ming Z, Liu X, Matsushita M, Fujita T. Specific binding of L-ficolin and H-ficolin to apoptotic cells leads to complement activation. Immunobiology. 2005;209(9):689-97. doi: 10.1016/j.imbio.2004.11.001. PMID 15804047
- [Background] Herrmann M, Voll RE, Zoller OM, Hagenhofer M, Ponner BB, Kalden JR. Impaired phagocytosis of apoptotic cell material by monocyte-derived macrophages from patients with systemic lupus erythematosus. Arthritis Rheum. 1998 Jul;41(7):1241-50. doi: 10.1002/1529-0131(199807)41:73.0.CO;2-H. PMID 9663482
- [Background] Liphaus BL, Kiss MH. The role of apoptosis proteins and complement components in the etiopathogenesis of systemic lupus erythematosus. Clinics (Sao Paulo). 2010 Mar;65(3):327-33. doi: 10.1590/S1807-59322010000300014. PMID 20360925
- [Background] Orbai AM, Truedsson L, Sturfelt G, Nived O, Fang H, Alarcon GS, Gordon C, Merrill J, Fortin PR, Bruce IN, Isenberg DA, Wallace DJ, Ramsey-Goldman R, Bae SC, Hanly JG, Sanchez-Guerrero J, Clarke AE, Aranow CB, Manzi S, Urowitz MB, Gladman DD, Kalunian KC, Costner MI, Werth VP, Zoma A, Bernatsky S, Ruiz-Irastorza G, Khamashta MA, Jacobsen S, Buyon JP, Maddison P, Dooley MA, Van Vollenhoven RF, Ginzler E, Stoll T, Peschken C, Jorizzo JL, Callen JP, Lim SS, Fessler BJ, Inanc M, Kamen DL, Rahman A, Steinsson K, Franks AG Jr, Sigler L, Hameed S, Pham N, Brey R, Weisman MH, McGwin G Jr, Magder LS, Petri M. Anti-C1q antibodies in systemic lupus erythematosus. Lupus. 2015 Jan;24(1):42-9. doi: 10.1177/0961203314547791. Epub 2014 Aug 14. PMID 25124676
- [Background] Sato N, Ohsawa I, Nagamachi S, Ishii M, Kusaba G, Inoshita H, Toki A, Horikoshi S, Ohi H, Matsushita M, Tomino Y. Significance of glomerular activation of the alternative pathway and lectin pathway in lupus nephritis. Lupus. 2011 Nov;20(13):1378-86. doi: 10.1177/0961203311415561. Epub 2011 Sep 5. PMID 21893562
- [Background] Lacroix M, Dumestre-Perard C, Schoehn G, Houen G, Cesbron JY, Arlaud GJ, Thielens NM. Residue Lys57 in the collagen-like region of human L-ficolin and its counterpart Lys47 in H-ficolin play a key role in the interaction with the mannan-binding lectin-associated serine proteases and the collectin receptor calreticulin. J Immunol. 2009 Jan 1;182(1):456-65. doi: 10.4049/jimmunol.182.1.456. PMID 19109177
- [Background] Plawecki M, Lheritier E, Clavarino G, Jourde-Chiche N, Ouili S, Paul S, Gout E, Sarrot-Reynauld F, Bardin N, Boelle PY, Chiche L, Bouillet L, Thielens NM, Cesbron JY, Dumestre-Perard C. Association between the Presence of Autoantibodies Targeting Ficolin-3 and Active Nephritis in Patients with Systemic Lupus Erythematosus. PLoS One. 2016 Sep 15;11(9):e0160879. doi: 10.1371/journal.pone.0160879. eCollection 2016. PMID 27631981
- [Background] Tanha N, Pilely K, Faurschou M, Garred P, Jacobsen S. Plasma ficolin levels and risk of nephritis in Danish patients with systemic lupus erythematosus. Clin Rheumatol. 2017 Feb;36(2):335-341. doi: 10.1007/s10067-016-3508-2. Epub 2016 Dec 15. PMID 27981461
- [Background] Watanabe H, Saito R, Asano T, Sato S, Iwadate H, Kobayashi H, Ohira H. Serum L-ficolin levels in patients with systemic lupus erythematosus. Mod Rheumatol. 2012 Nov;22(6):899-902. doi: 10.1007/s10165-012-0616-y. Epub 2012 Feb 21. PMID 22350641
- [Derived] Colliard S, Jourde-Chiche N, Clavarino G, Sarrot-Reynauld F, Gout E, Deroux A, Fougere M, Bardin N, Bouillet L, Cesbron JY, Thielens NM, Dumestre-Perard C. Autoantibodies Targeting Ficolin-2 in Systemic Lupus Erythematosus Patients With Active Nephritis. Arthritis Care Res (Hoboken). 2018 Aug;70(8):1263-1268. doi: 10.1002/acr.23449. Epub 2018 Jun 21. PMID 29045037